CLINICAL TRIAL: NCT05883891
Title: Prothrombin Time Predicts Steroid Response in Severe Alcoholic Hepatitis.
Acronym: AH2023
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5840
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Alcoholic Hepatitis
Keywords: early liver transplantation; alcohol; cirrhosis; corticosteroid therapy; Maddrey's discriminant function; Lille score; prothrombin time; Alcohol Use Disorder; steroid response
MeSH Terms: conditions — Hepatitis, Alcoholic; Fibrosis; Alcoholism | interventions — Prothrombin Time

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe alcoholic hepatitis: Patients admitted with a clinical diagnosis of severe alcoholic hepatitis eligible to corticosteroid treatment. Prothrombin time at diagnosis was registered to evaluate wether it correlated with Lille score at day 7 and therefore response to standard medical treatment.
  Interventions: Diagnostic Test: prothrombin time

INTERVENTIONS:
Diagnostic Test: prothrombin time — Prothrombin time at value at diagnosis was used to assess the presence of a correlation with Lille score at day 7 and therefore wether it could predict response to medical treatment.

SUMMARY:
Alcoholic hepatitis (AH) is the most severe form of acute alcohol-related liver disease. Maddrey's discriminant function (mDF) >32 defines the severe form of AH, which is associated with a high mortality. Corticosteroid therapy (CS) represents the main medical treatment that may reduce short-term mortality. Lille score at day 7 assesses the therapeutic response to steroid therapy. At present, no parameters able to predict the response to steroid therapy have been highlighted. The mDF depends mainly on prothrombin time (PT). Aim of the present study was to evaluate if the PT value could predict the response to CS in severe AH (sAH).

ELIGIBILITY:
Inclusion Criteria:

- clinical diagnosis of first episode of severe alcoholic hepatitis with Maddrey's function score of 32 or higher, and the absence of contraindication to CS therapy (non-controlled infections/sepsis, hepatic encephalopathy, recent acute gastrointestinal bleeding, severe kidney dysfunction). The diagnosis of AH was based on the criteria of the National Institute on Alcohol Abuse and Alcoholism (NIAAA)-funded Alcoholic Hepatitis Consortia (Crabb DW, 2016). In particular, were enrolled in the study patients with: heavy alcohol use for >6 months, with an average consumption of more than 3 drinks (∼40 g) per day for women and 4 drinks (∼50-60 g) per day for men and with <30 days of abstinence before the onset of jaundice; AST/ALT ratio > 1.5 with an AST level > 45 IU/L (1.5 times upper limit of normal) and < 400 IU/L; serum bilirubin >3 mg/dL.

Exclusion Criteria:

* acute or chronic viral hepatitis,
* nonalcoholic steatohepatitis,
* cocaine use,
* drug-induced liver injury,
* fulminant Wilsons disease,
* hepatocellular carcinoma,
* portal vein thrombosis,
* biliary obstruction,
* severe autoimmune liver disease,
* neoplasms,
* severe comorbidities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Internal Medicine and Alcohol Related Diseases Unit of a teaching hospital with a clinical diagnosis of severe alcoholic hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
response to steroid treatment | seven days
  response to standard medical treatment assessed with Lille scoremat day 7

SECONDARY OUTCOMES:
death | 28 days
  death occurring during hospitalization from any cause
early liver transplantation | 7 days
  early transplantation in case of failure of medical treatment
infection | 28 days
  occurrence of opportunistic infections following steroid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Addolorato, Principal Investigator — Internal Medicine and Alcohol Related Disease Unit, Department of Medical and Surgical Sciences, Columbus-Gemelli Hospital, Fondazione Policlinico Universitario A. Gemelli IRCCS, Catholic University of Rome, Rome, Italy
Locations (1):
- Agostino Gemelli Polyclinic, Rome, Roma (provincia), Italy

IPD SHARING:
Plan to Share IPD: No